CLINICAL TRIAL: NCT00678600
Title: Optimizing HIV Disease-Specific Provider Alerts: A Randomized Controlled Informatics Trial Comparing Electronic Health Record (EHR) vs. Non-EHR Provider Alerts
Brief Title: Study of Provider Computer Alerts Designed to Improve Delivery of HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1K01AI062435 (NIH); K01AI062435 (NIH)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Informatics; Alerts; Toxicity; Virologic failure; Suboptimal follow up
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (static) Computer Alerts (Active Comparator): Participants in this arm will be assigned to standard care. Participants will be monitored for new laboratory toxicity, suboptimal follow up, and virologic failure. Provider computer alerts will be posted on the participant's electronic health record summary page.
  Interventions: Other: Standard (static) Computer Alerts
- Enhanced Computer Alerts (Experimental): Participants in this arm will be assigned to the enhanced alert arm. Participants will be monitored for new laboratory toxicity, suboptimal follow up, and virologic failure. Providers will receive population and asynchronous computer alerts with improved functionality.
  Interventions: Other: Enhanced Computer Alerts

INTERVENTIONS:
Other: Standard (static) Computer Alerts — Static Computer Alerts on Patient's EMR webpage.
  Arms: Standard (static) Computer Alerts
Other: Enhanced Computer Alerts — Population level and asynchronous alerts with enhanced functionality
  Arms: Enhanced Computer Alerts

SUMMARY:
The purpose of this study is to determine whether alerts independent of the ambulatory health record are more effective in eliciting physician responses and therefore have greater impact on HIV disease outcomes than traditional static alerts.

DETAILED DESCRIPTION:
This study will compare the effectiveness of standard and enhanced care alerts in HIV infected participants at Massachusetts General Hospital in Boston, Massachusetts.

Participants will be a part of this study for 4 years or until they are no longer followed at Massachusetts General Hospital. Participants will be assigned randomly to one of two arms. Participants assigned to Arm 1 will receive standard care, involving standard provider alerts which will be posted on the participant's health record. Participants assigned to Arm 2 will receive enhanced care, involving improved functionality. Experimental informatics-based provider alerts and support systems will be used to develop a pilot system designed to optimize delivery of HIV clinical care.

All participants will be monitored for new laboratory toxicities, suboptimal follow up, and virologic failure at their normally scheduled appointments.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Followed in the Massachusetts General Hospital HIV clinic.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in CD4 count | Throughout study

SECONDARY OUTCOMES:
Time to repeat laboratory testing | Throughout study
Time to follow up appointment | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Robbins, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Robbins GK, Lester W, Johnson KL, Chang Y, Estey G, Surrao D, Zachary K, Lammert SM, Chueh HC, Meigs JB, Freedberg KA. Efficacy of a clinical decision-support system in an HIV practice: a randomized trial. Ann Intern Med. 2012 Dec 4;157(11):757-66. doi: 10.7326/0003-4819-157-11-201212040-00003. PMID 23208165